CLINICAL TRIAL: NCT03723642
Title: Investigation of Oxidative Stress - Open Appendectomy (OAE) Versus Laparoscopic Appendectomy (LAE) in Childhood and Adolescence - A Pilot Study
Brief Title: Investigation of Oxidative Stress in Appendectomy - Open Versus Laparoscopic in Childhood and Adolescence
Acronym: OSAE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Graz (Other)
Collaborators: University of Rostock (Other); Graz University of Technology (Other)
Responsible Party: Principal Investigator, Warncke Gert, MD, Principal Investigator, Medical University of Graz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 30-120 ex 17/18
Record Dates: First submitted 2018-07-10; First posted 2018-10-29 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Appendicitis Acute
Keywords: acute appendicitis; volatile organic compounds; oxidative stress; laparoscopic appendectomy; open appendectomy
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Intervention Model Description: 40 patients aged 6-18 years suffering from acute appendicitis are to be included. These are divided into 2 groups. Group 1 (n = 20) with laparoscopic and group 2 (n = 20) with open appendectomy.
Who Masked: Participant
Masking Description: After obtaining written informed consent from patients/legal guardians the patients will be randomized 1:1 to one of the two surgical techniques. Randomization is carried out using the web-based "Randomizer for Clinical Trials" program at the Institute of Medical Informatics, Statistics and Documentation at the Medical University of Graz (www.randomizer.at).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OAE group (Active Comparator): All patients will undergo measurements of oxydative stress (initial serum malondialdehyde level and final serum malondialdehyde level), White blood cell count (initial differential white blood cell count and final differential white blood cell count), c-reactive protein measurements (initial c-reactive protein serum level and final c-reactive protein serum level) as well as volatile organic compound (VOC) sampling (initial VOC, VOC 5min, VOC 15min, VOC 30min, VOC 45min and final VOC).
  Interventions: Diagnostic Test: Initial serum malondialdehyde level; Diagnostic Test: Final serum malondialdehyde level; Diagnostic Test: Initial differential white blood cell count; Diagnostic Test: Final differential white blood cell count; Diagnostic Test: Initial c-reactive protein serum level; Diagnostic Test: Final c-reactive protein serum level; Diagnostic Test: Initial VOC; Diagnostic Test: VOC 5min; Diagnostic Test: VOC 15min; Diagnostic Test: VOC 30min; Diagnostic Test: VOC 45min; Diagnostic Test: Final VOC
- LAE group (Active Comparator): All patients will undergo measurements of oxydative stress (initial serum malondialdehyde level and final serum malondialdehyde level), White blood cell count (initial differential white blood cell count and final differential white blood cell count), c-reactive protein measurements (initial c-reactive protein serum level and final c-reactive protein serum level) as well as volatile organic compound (VOC) sampling (initial VOC, VOC 5min, VOC 15min, VOC 30min, VOC 45min and final VOC).
  Interventions: Diagnostic Test: Initial serum malondialdehyde level; Diagnostic Test: Final serum malondialdehyde level; Diagnostic Test: Initial differential white blood cell count; Diagnostic Test: Final differential white blood cell count; Diagnostic Test: Initial c-reactive protein serum level; Diagnostic Test: Final c-reactive protein serum level; Diagnostic Test: Initial VOC; Diagnostic Test: VOC 5min; Diagnostic Test: VOC 15min; Diagnostic Test: VOC 30min; Diagnostic Test: VOC 45min; Diagnostic Test: Final VOC

INTERVENTIONS:
Diagnostic Test: Initial serum malondialdehyde level — Blood sample (0.4ml) will be obtained within 5 minutes before induction of general anaesthesia.
  Samples will be obtained in both groups (LAE and OAE)
Diagnostic Test: Final serum malondialdehyde level — Blood sample (0.4ml) will be obtained within 5 minutes after wound closure. Samples will be obtained in both groups (LAE and OAE)
Diagnostic Test: Initial differential white blood cell count — Differential blood counts (microscopic) will be obtained during pre-operative routine work-up.
  Samples will be obtained in both groups (LAE and OAE).
Diagnostic Test: Final differential white blood cell count — Differential blood counts (microscopic) will be obtained 24h after the first sample (Initial differential blood count).
  Samples will be obtained in both groups (LAE and OAE).
Diagnostic Test: Initial c-reactive protein serum level — C-reactive protein levels will be obtained during pre-operative routine work-up.
  Samples will be obtained in both groups (LAE and OAE).
Diagnostic Test: Final c-reactive protein serum level — C-reactive protein levels will be obtained 24h after the first sample (initial c-reactive protein level).
  Samples will be obtained in both groups (LAE and OAE).
Diagnostic Test: Initial VOC — Volatile organic compound sampling (2 samples within 5 minutes) within 10 minutes before induction of general anesthesia
Diagnostic Test: VOC 5min — Volatile organic compound sampling (2 samples within5 minutes) within 5 minutes after endotracheal intubation before skin incision.
Diagnostic Test: VOC 15min — Volatile organic compound sampling (2 samples within 5 minutes) 15 minutes after skin incision.
Diagnostic Test: VOC 30min — Volatile organic compound sampling (2 samples within 5 minutes) 30 minutes after skin incision.
Diagnostic Test: VOC 45min — Volatile organic compound sampling (2 samples within 5 minutes) 45 minutes after skin incision.
Diagnostic Test: Final VOC — Volatile organic compound sampling (2 samples within 5 minutes) within 5 minutes after skin closure.

SUMMARY:
In the planned prospective randomized study, oxidative stress will be investigated by analyzing volatile organic compounds in the exhaled air in children. Children who have undergone open versus laparoscopic surgery for appendicitis will be compared. A better understanding of the effects of the surgical technique could be a prerequisite for an optimized surgical setting. It could also lead to recommendations for pre- or perioperatively antioxidative agents.

DETAILED DESCRIPTION:
Aim of the study: In the planned prospective randomized study, oxidative stress will be investigated by analyzing VOCs (volatile organic compounds) in the exhaled breath in children undergoing open or laparoscopic surgery for appendicitis at the Department of Pediatric and Adolescent Surgery of the Medical University of Graz. A resulting better understanding of the effects of the surgical technique can a) be a pre-condition for an optimized surgical setting and b) possibly lead to recommendations of pre- or perioperatively antioxidatively active substances and c) be a base for future surgical procedures.

Study design: This is a prospective randomized pilot study in children and adolescents undergoing surgery due to acute appendicitis. Patients with complicated appendicitis and those with an intraoperatively caused disorder will be excluded. The operation within the context of this study is exclusively conducted by specialists of the Department of Pediatric and Adolescent Surgery of the Medical University of Graz, who perform both - open and laparoscopic surgical techniques. 40 patients aged 6-18 years suffering from acute appendicitis are to be included. These are divided into 2 groups. Group 1 (n = 20) with laparoscopic and group 2 (n = 20) with open appendectomy.

Recruitment and compensation of study participants: Parents/patients are made aware of the study by means of an information sheet and are provided with a declaration of consent if interested. Participants do not receive any compensation for participating in the study.

Sampling of exhaled VOCs (volatile organic compounds) using NTME (needle trap microextraction) for measurement OS (oxidative stress): Number of samples: 2 samples each from exhaled breath at the times defined below (in total n = 12). The time of sampling: t1 before anaesthetic introduction (n = 2); t2 after anesthetic introduction (n = 2); t3 15 minutes after cut (n = 2); t4 30 minutes after cut (n = 2); t5 45 minutes after cut (n = 2); t6 after seam (n = 2).

Analysis of exhaled VOCs for measurement OS: The exhaled breath samples taken are placed in an injector of a gas chromatograph into the inert carrier gas stream (He). The substances are assigned according to their retention time in the chromatogram and its mass spectrum. Unknown connections in the mass spectrum of exhaled breath is used as a basis for comparison with a reference database.

Sampling of blood markers for measurement OS: a) sampling times for WBCs, CRP: t1 = 1 sample preoperatively (before anaesthetic introduction) and t2 = 1 sample after 24 h. b) sampling times for malondialdehyde: t1 = 1 sample before anaesthetic introduction and t2 = 1 sample after suture.

Histopathological grading: The explanted vermiform appendix becomes the histopathological Refurbishment at the Institute of Pathology of the Medical University of Graz. There the classification is made according to the histopathological findings in 4 degrees of severity (acute focal appendicitis, acute suppurative appendicitis, acut gangrenous appendicitis, perforated appendicitis).

Sampling WBCs, CRP: These are carried out within the scope of routine diagnostics due to the clinical presentation of the AA (acute appendicitis).

Sampling VOCs: 2 breath samples are taken from each patient during expiration, taken from it. To collect the samples, the investigators use an automatic Sampling device connected directly to a capnometer. This system works with microextraction (NTME) and enables a automatic sampling of the alveolar air, i.e. in the plateau of the CO2 curve. The samples are sent to the Intitute of Rostock Medical Breath Analysis and Technologies (RoMBAT) as cooperation partner. This partner was selected because it already has extensive experience with the methodology and studies on oxidative stress during operations.

Malondialdehyde (MDA) sampling: Malondialdehyde is analysed at the Clinical Institute for Medical and Chemical Laboratory Diagnostics at the Medical University of Graz means of ultra-modern GC-MS method. For this purpose, the patient is assigned to the two Measuring times 2 x 400 μl EDTA plasma taken. The second sample serves only as a safety measure if repeat measurements are necessary. The samples obtained must be deep-frozen at -80 °C within 2 hours. . Subsequently (at the latest on the following day) the samples must be analyzed to the Institute.

Planned evaluation: The statistical investigations are carried out with SPSS 23.0®. Graphical representation of the data is performed with GraphPad Prism 7®. To investigate whether the main target variables (VOCs) differ in the course between the two groups, linear models are used for repeated measurements with group (open versus laparoscopic appendectomy) as intermediate subject factor and time of measurement (t1 to t6) as internal subject factor. In the case of deviations from the normal distribution, transformations are taken into consideration. The secondary targets, i.e. the changes in the serum markers on theTimes t1 and t6, are compared between the 2 groups (open versus laparoscopic appendectomy) by Mann-Whitney U-test (data not normally distributed) or independent T-test (with normal distribution). In order to establish relationships between the VOCs and the serum markers for oxidative stress at times t1 and t6 a correlation analysis is performed (depending on the data, Pearson or Spearman Rho). All statistical tests are carried out on two sides and all p-values are interpreted purely exploratively.

ELIGIBILITY:
Inclusion Criteria:

* Age from 6-18 years
* reliable diagnosis of acute appendicitis
* surgical therapy using open/laparoscopic surgical technique
* given approval

Exclusion Criteria:

* Age not between 6 and 18 years
* chronic underlying disease/autoimmune disease
* complicated appendicitis (perforation, consecutive purulent peritonitis, abscess formation)
* infection outside acute appendicitis
* SIRS
* taking medications containing the cytochrome P450 (CYP) system affect including cortisone
* impaired liver function
* unaccepted consent

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-10-02 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Are volatile respiratory gas markers for oxidative stress (such as pentanes, isoprenes) dependent on the surgical method (open versus laparoscopic appendectomy)? | 1 year
  We investigate the respiratory volatile organic compounds before, during and at the end of surgery and compare the respiratory gas profiles of the two groups open versus laparoscopic appendectomy.

SECONDARY OUTCOMES:
Alterations of serum malondialdehyde serum levels. | 1 year
  The changes of the serum marker for oxidative stress MDH before and after surgery will be investigated and the changes in open versus laparoscopic appendectomy will be compared. One sample will be taken preoperatively and one sample postoperatively.
Alterations of inflammation markers. | 1 year
  The changes of the serum inflammation markers before and after surgery will be investigated and the changes in open versus laparoscopic appendectomy will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Holger Till, MD, Study Director — Department of Pediatric and Adolescent Surgery, Medical University of Graz; Gert Warncke, MD, Principal Investigator — Department of Pediatric and Adolescent Medicine, Medical University of Graz
Locations (1):
- Department of Paediatric and Adolescent Surgery, Graz, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stringer MD. Acute appendicitis. J Paediatr Child Health. 2017 Nov;53(11):1071-1076. doi: 10.1111/jpc.13737. Epub 2017 Oct 17. PMID 29044790
- [Background] Ohmann C, Franke C, Kraemer M, Yang Q. [Status report on epidemiology of acute appendicitis]. Chirurg. 2002 Aug;73(8):769-76. doi: 10.1007/s00104-002-0512-7. German. PMID 12425152
- [Background] Gorter RR, Eker HH, Gorter-Stam MA, Abis GS, Acharya A, Ankersmit M, Antoniou SA, Arolfo S, Babic B, Boni L, Bruntink M, van Dam DA, Defoort B, Deijen CL, DeLacy FB, Go PM, Harmsen AM, van den Helder RS, Iordache F, Ket JC, Muysoms FE, Ozmen MM, Papoulas M, Rhodes M, Straatman J, Tenhagen M, Turrado V, Vereczkei A, Vilallonga R, Deelder JD, Bonjer J. Diagnosis and management of acute appendicitis. EAES consensus development conference 2015. Surg Endosc. 2016 Nov;30(11):4668-4690. doi: 10.1007/s00464-016-5245-7. Epub 2016 Sep 22. PMID 27660247
- [Background] Binnebosel M, Otto J, Stumpf M, Mahnken AH, Gassler N, Schumpelick V, Truong S. [Acute appendicitis. Modern diagnostics--surgical ultrasound]. Chirurg. 2009 Jul;80(7):579-87. doi: 10.1007/s00104-009-1684-1. German. PMID 19471900
- [Background] Kim M, Kim SJ, Cho HJ. International normalized ratio and serum C-reactive protein are feasible markers to predict complicated appendicitis. World J Emerg Surg. 2016 Jun 21;11:31. doi: 10.1186/s13017-016-0081-6. eCollection 2016. PMID 27330547
- [Background] Svensson JF, Hall NJ, Eaton S, Pierro A, Wester T. A review of conservative treatment of acute appendicitis. Eur J Pediatr Surg. 2012 Jun;22(3):185-94. doi: 10.1055/s-0032-1320014. Epub 2012 Jul 5. PMID 22767171
- [Background] Blakely ML, Williams R, Dassinger MS, Eubanks JW 3rd, Fischer P, Huang EY, Paton E, Culbreath B, Hester A, Streck C, Hixson SD, Langham MR Jr. Early vs interval appendectomy for children with perforated appendicitis. Arch Surg. 2011 Jun;146(6):660-5. doi: 10.1001/archsurg.2011.6. Epub 2011 Feb 21. PMID 21339413
- [Background] Whyte C, Levin T, Harris BH. Early decisions in perforated appendicitis in children: lessons from a study of nonoperative management. J Pediatr Surg. 2008 Aug;43(8):1459-63. doi: 10.1016/j.jpedsurg.2007.11.032. PMID 18675635
- [Background] Li X, Zhang J, Sang L, Zhang W, Chu Z, Li X, Liu Y. Laparoscopic versus conventional appendectomy--a meta-analysis of randomized controlled trials. BMC Gastroenterol. 2010 Nov 3;10:129. doi: 10.1186/1471-230X-10-129. PMID 21047410
- [Background] Coccolini F, Trana C, Sartelli M, Catena F, Di Saverio S, Manfredi R, Montori G, Ceresoli M, Falcone C, Ansaloni L. Laparoscopic management of intra-abdominal infections: Systematic review of the literature. World J Gastrointest Surg. 2015 Aug 27;7(8):160-9. doi: 10.4240/wjgs.v7.i8.160. PMID 26328036
- [Background] Ciftci F. Laparoscopic vs mini-incision open appendectomy. World J Gastrointest Surg. 2015 Oct 27;7(10):267-72. doi: 10.4240/wjgs.v7.i10.267. PMID 26525039
- [Background] Noviello C, Romano M, Martino A, Cobellis G. Transumbilical Laparoscopic-Assisted Appendectomy in the Treatment of Acute Uncomplicated Appendicitis in Children. Gastroenterol Res Pract. 2015;2015:949162. doi: 10.1155/2015/949162. Epub 2015 Sep 29. PMID 26491433
- [Background] Khan SY, Al-Balushi ZN, Bhatti KM, Ehsan T, Mandhan P. Cost Comparison between Laparoscopic and Open Appendectomies in Children. Sultan Qaboos Univ Med J. 2013 May;13(2):275-9. doi: 10.12816/0003234. Epub 2013 May 9. PMID 23862034
- [Background] Zelzer S, Oberreither R, Bernecker C, Stelzer I, Truschnig-Wilders M, Fauler G. Measurement of total and free malondialdehyde by gas-chromatography mass spectrometry--comparison with high-performance liquid chromatography methology. Free Radic Res. 2013 Aug;47(8):651-6. doi: 10.3109/10715762.2013.812205. Epub 2013 Jul 2. PMID 23745592
- [Background] McCrum-Gardner E. Which is the correct statistical test to use? Br J Oral Maxillofac Surg. 2008 Jan;46(1):38-41. doi: 10.1016/j.bjoms.2007.09.002. Epub 2007 Oct 24. PMID 17961892
- [Result] Kapischke M, Pries A, Caliebe A. Short term and long term results after open vs. laparoscopic appendectomy in childhood and adolescence: a subgroup analysis. BMC Pediatr. 2013 Oct 1;13:154. doi: 10.1186/1471-2431-13-154. PMID 24079822
- [Result] Jaschinski T, Mosch C, Eikermann M, Neugebauer EA. Laparoscopic versus open appendectomy in patients with suspected appendicitis: a systematic review of meta-analyses of randomised controlled trials. BMC Gastroenterol. 2015 Apr 15;15:48. doi: 10.1186/s12876-015-0277-3. PMID 25884671
- [Result] Minutolo V, Licciardello A, Di Stefano B, Arena M, Arena G, Antonacci V. Outcomes and cost analysis of laparoscopic versus open appendectomy for treatment of acute appendicitis: 4-years experience in a district hospital. BMC Surg. 2014 Mar 19;14:14. doi: 10.1186/1471-2482-14-14. PMID 24646120
- [Result] Tsai CC, Lee SY, Huang FC. Laparoscopic versus open appendectomy in the management of all stages of acute appendicitis in children: a retrospective study. Pediatr Neonatol. 2012 Oct;53(5):289-94. doi: 10.1016/j.pedneo.2012.07.002. Epub 2012 Sep 1. PMID 23084720
- [Result] Stipancic I, Zarkovic N, Servis D, Sabolovic S, Tatzber F, Busic Z. Oxidative stress markers after laparoscopic and open cholecystectomy. J Laparoendosc Adv Surg Tech A. 2005 Aug;15(4):347-52. doi: 10.1089/lap.2005.15.347. PMID 16108734
- [Result] Jakimowicz J, Stultiens G, Smulders F. Laparoscopic insufflation of the abdomen reduces portal venous flow. Surg Endosc. 1998 Feb;12(2):129-32. doi: 10.1007/s004649900612. PMID 9479726
- [Result] Baysal Z, Togrul T, Aksoy N, Cengiz M, Celik H, Boleken ME, Kaya M, Yavuz G. Evaluation of total oxidative and antioxidative status in pediatric patients undergoing laparoscopic surgery. J Pediatr Surg. 2009 Jul;44(7):1367-70. doi: 10.1016/j.jpedsurg.2008.11.031. PMID 19573663
- [Result] Aktimur R, Gokakin AK, Deveci K, Atabey M, Topcu O. Oxidative stress markers in laparoscopic vs. open appendectomy for acute appendicitis: A double-blind randomized study. J Minim Access Surg. 2016 Apr-Jun;12(2):143-7. doi: 10.4103/0972-9941.156203. PMID 27073307
- [Result] Schubert JK, Miekisch W, Geiger K, Noldge-Schomburg GF. Breath analysis in critically ill patients: potential and limitations. Expert Rev Mol Diagn. 2004 Sep;4(5):619-29. doi: 10.1586/14737159.4.5.619. PMID 15347256
- [Result] Miekisch W, Schubert JK, Noeldge-Schomburg GF. Diagnostic potential of breath analysis--focus on volatile organic compounds. Clin Chim Acta. 2004 Sep;347(1-2):25-39. doi: 10.1016/j.cccn.2004.04.023. PMID 15313139
- [Result] Pabst F, Miekisch W, Fuchs P, Kischkel S, Schubert JK. Monitoring of oxidative and metabolic stress during cardiac surgery by means of breath biomarkers: an observational study. J Cardiothorac Surg. 2007 Sep 18;2:37. doi: 10.1186/1749-8090-2-37. PMID 17877828
- [Result] Trefz P, Rosner L, Hein D, Schubert JK, Miekisch W. Evaluation of needle trap micro-extraction and automatic alveolar sampling for point-of-care breath analysis. Anal Bioanal Chem. 2013 Apr;405(10):3105-15. doi: 10.1007/s00216-013-6781-9. Epub 2013 Feb 7. PMID 23388692